CLINICAL TRIAL: NCT02835183
Title: Prospective Evaluation of iDECIDE: A Smartphone App for Insulin Bolus Dosing
Brief Title: Evaluation of iDECIDE: A Smartphone App for Insulin Dosing Accounting for Alcohol and Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adela Grando, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: iDECIDEEvaluation
Record Dates: First submitted 2016-06-06; First posted 2016-07-15 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin pump followed by iDECIDE (Experimental): Participants will be randomly assigned to 4 weeks of using their insulin pump to decide insulin boluses and then 4 weeks of using iDECIDE to receive recommendations for insulin dosing.
  Interventions: Device: iDECIDE; Device: Insulin pump
- iDECIDE followed by insulin pump (Experimental): Participants will be randomly assigned to 4 weeks of using iDECIDE to receive recommendations for insulin dosing and then 4 weeks of using their insulin pump to decide insulin boluses.
  Interventions: Device: iDECIDE; Device: Insulin pump

INTERVENTIONS:
Device: iDECIDE — The iDECIDE app will be installed in study participant's smartphone. The app requests from study participants input on food consumed (included food's carbohydrate content), alcohol consumed (included alcohol's carbohydrate content) and exercise plans (including duration and intensity). Based on that input the app suggests insulin bolus dosing.
Device: Insulin pump — Study participants will use during the study their own insulin pump and continuous glucose sensor. As inclusion criteria, investigators expect study participants to have been using their insulin pump and continuous glucose sensor for at least one year.

SUMMARY:
The investigators propose a randomized cross-over study Phase 1 Clinical trial. 30 type 1 diabetes adult outpatients using insulin pumps and continuous glucose monitoring system will be recruited from the Endocrinology Clinic at the Mayo Clinic Arizona. Participants will be randomly assigned to 4 weeks of using their pump bolus wizards to decide insulin boluses and then 4 wks of using iDECIDE to receive recommendations for insulin dosing, or vice versa. The primary outcomes to compare iDECIDE's insulin dosing algorithm against the pump calculators will be: mean postprandial glucose level and number of events with excessive blood glucose highs and lows.

DETAILED DESCRIPTION:
The investigators will seek approval from Mayo Clinic and Arizona State University Institutional Review Board to recruit 30 type 1 diabetes adult outpatients using insulin pumps and continuous glucose monitoring system from the Endocrinology Clinic at Mayo Clinic Arizona. First, participants will complete a questionnaire to self-assess their confidence to count carbs from food/drinks, personal perceptions on how exercise/alcohol affect their blood glucose, and how they learned about it (e.g., trial and error, education from providers), and compensation techniques used to adjust for exercise performed/alcohol consumed (for instance, adjust for basal rate or adjust insulin boluses). Stored glucose data will be analyzed for the previous 8 weeks prior to entry to establish patient-specific upper and lower bounds for determining excessive blood glucose highs and lows. Second, participants will be randomly assigned to 4 weeks of using their pump bolus wizards to decide insulin boluses and then 4 weeks of using iDECIDE to receive recommendations for insulin dosing, or vice versa. Throughout the 8 weeks, study participants will be asked to wear a wristband heart rate accelerometer that will provide data on time and duration of exercise performed. Also, during the 8 weeks, study participants will use their glucose sensor and pump to measure blood glucose and to deliver basal insulin. During the 4 weeks when participants receive recommendations from iDECIDE, the pump's bolus calculator will be turned off so participants will receive no insulin bolus recommendations from pump. While receiving recommendations from iDECIDE, participants will use the pump to manually deliver insulin boluses and can either use the advice from iDECIDE or override it.

The primary outcomes to compare iDECIDE's insulin dosing algorithm against the pump calculators will be: mean postprandial glucose level and number of events with excessive blood glucose highs and lows. Potential secondary outcomes: mean percentage of time with low glucose level and time spent in the target glucose range.

ELIGIBILITY:
Inclusion Criteria:

* Mayo Clinic Arizona type 1 diabetes outpatients,
* Older than 18 years and younger than 60,
* Non-pregnant,
* English speakers,
* Who use Medtronic insulin pumps and continuous glucose monitoring sensors,
* Own a smartphone,
* Have kept in consistent contact with the Mayo Clinic Division of Endocrinology health care team during the last year, and have use the same insulin pump and continuous glucose sensor for at least one year.

Exclusion Criteria:

* Subjects who do not satisfy the inclusion criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Compare mean postprandial glucose level | 2 months
  Compare iDECIDE's insulin dosing algorithm against the pump calculators in terms of mean postprandial glucose level

SECONDARY OUTCOMES:
Hypoglycemia events | 2 months
  % time with blood glucose < 3.9 mmol/L
Hyperglycemia events | 2 months
  % time with blood glucose > 8.0 mmol/L

IPD SHARING:
Plan to Share IPD: No